CLINICAL TRIAL: NCT01978080
Title: ETSense: Adaptive Portable Essential Tremor Monitor - Symptomatic Impact Study
Brief Title: Continuous Tremor Assessment During Daily Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: Rush University Medical Center (Other); Baylor College of Medicine (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5R44AG034708-03 (NIH); 5R44AG034708 (NIH)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Tremor reports provided (Experimental): Kinesia HomeView utilized to monitor tremor at home and reports provided to treating clinician
  Interventions: Device: Kinesia HomeView
- Tremor reports not provided (Active Comparator): Kinesia HomeView utilized to monitor tremor at home and reports not provided to treating clinician
  Interventions: Device: Kinesia HomeView

INTERVENTIONS:
Device: Kinesia HomeView

SUMMARY:
The specific aim of this study is to evaluate if tremor severity and quality of life can be improved more using continuous home monitoring along with traditional assessments versus traditional assessments alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with essential tremor
* Currently taking medication to control tremor

Exclusion Criteria:

* Cognitive limitations that prevent comprehension or execution of study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Change Scale score | End of Month 1, End of Month 2, End of Month 3
  Utilized to measure any improvement or worsening of symptoms relative to a baseline state at enrollment

SECONDARY OUTCOMES:
Clinical Global Impression-Severity Scale Score | Enrollment, End of Month 1, End of Month 2, End of Month 3
  Utilized to measure overall tremor severity
Washington Heights Inwood Genetic Study of Essential Tremor (WHIGET) Tremor Rating Scale | Enrollment, End of Month 1, End of Month 2, End of Month 3
  Utilized to measure overall tremor severity
Quality of Life in Essential Tremor Questionnaire | Enrollment, End of Month 1, End of Month 2, End of Month 3
  Utilized to measure the impact tremor has on overall quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Baylor College of Medicine, Houston, Texas